CLINICAL TRIAL: NCT03710278
Title: The Effectiveness and Safety of Human Lumbar Puncture Assist Device (LPat)
Acronym: LPat
Status: Completed | Type: Observational
Sponsor: Spartanburg Regional Healthcare System (Other)
Collaborators: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Hanna S. Sahhar, Medical Director, PICU, Spartanburg Regional Healthcare System
Other Study IDs: Pro00073159
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Meningitis; Encephalitis; Guillain-Barré; Subarachnoid Hemorrhage; Intracranial Neoplasm; Intracranial CNS Disorder
MeSH Terms: conditions — Meningitis; Encephalitis; Guillain-Barre Syndrome; Subarachnoid Hemorrhage; Brain Neoplasms; Brain Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- LPat Device: Performing Lumbar Puncture assisted by LPat
  Interventions: Device: LPat Device

INTERVENTIONS:
Device: LPat Device — Performing Lumbar Puncture utilizing LPat device
  Other Names: Lumbar Puncture Assisted by LPat

SUMMARY:
The purpose of this study is to proof and investigate the effectiveness and safety of the invented device named "Human Lumbar Puncture Assist Device (LPat)" as an assist tool to be utilized to improve the success rate of performing lumbar puncture (LP), avoid side effects from multiple punctures, avoid excess radiation if the LP need to be done under fluoroscopy, and need to obtain none traumatic tap for better CSF analysis.

DETAILED DESCRIPTION:
"Human Lumbar Puncture Assist Device (LPat)" was invented as an assist tool to be utilized to improve the success rate of performing lumbar puncture (LP), avoid side effects from multiple punctures, avoid excess radiation.

ELIGIBILITY:
Inclusion Criteria:

Patients age 12 years and older who need lumbar puncture (LP) for diagnostic purposes or patients already underwent LP but failed to obtain Cerebrospinal Fluids i.e. "Unsuccessful Tap"

Exclusion Criteria:

Patients younger than 12 years of age

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient 12 years or older
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Successful Lumbar Puncture | Immediate
  Obtain CSF

CONTACTS AND LOCATIONS:
Locations (1):
- Spartanburg Reginal Heathcare System, Spartanburg, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No